CLINICAL TRIAL: NCT01042951
Title: Randomized, Double-blind, Placebo-controlled Trial, to Evaluate the Safety and Immunogenicity of Orally Administered, Killed, Bivalent Whole-cell, Cholera Vaccine, ShanChol in Bangladeshi Adults and Children
Brief Title: To Determine the Safety and Immunogenicity of an Oral Whole Cell ShanChol Cholera Vaccine in Bangladesh
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: International Centre for Diarrhoeal Disease Research, Bangladesh (Other)
Collaborators: International Vaccine Institute (Other); Government of Bangladesh (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: PR-09047
Record Dates: First submitted 2010-01-05; First posted 2010-01-06 (Estimated); Last update posted 2014-10-30 (Estimated); Status verified 2010-01

CONDITIONS: Healthy
Keywords: safety; immunogenicity; Healthy Participants

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ShanChol Cholera Vaccine (Active Comparator)
  Interventions: Biological: ShanChol Cholera Vaccine
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: ShanChol Cholera Vaccine — 55 adults (18-45 year old) will be given 2 doses of the bivalent whole-cell cholera vaccine 55 Toddlers(2-5 years) will be given 2 doses of the bivalent whole-cell cholera vaccine 55 Younger children(12-23 months)will be given 2 doses of the bivalent whole-cell cholera vaccine
  Other Names: ShanCholCholera Vaccine
  Arms: ShanChol Cholera Vaccine
Other: Placebo — 55 adults (18-45 year old) will be given 2 doses placebo, 55 Toddlers(2-5 years) will be given 2 doses of placebo, and 55 Younger children(12-23 months)will be given 2 doses of placebo
  Arms: Placebo

SUMMARY:
Background: Severe dehydrating cholera due to V. cholerae O1 is an important public health problem in Bangladesh and many other developing countries. V. cholerae O1 is a major bacterial pathogen causing around 5 million cases and at least 200,000 deaths in adults and children each year. It can be assumed that there are at least 300,000 severe cases and 1.2 million infections in people in Bangladesh alone. The rate of cholera varies from around 1 to 8 per 1000 population and the highest attack rate is in children 2- to 9-year years of age . Cholera is now also being documented in very young children. Currently enteric vaccine approaches are regarded as the most accessible short term and practical means to prevent and control such illnesses to prevent disease and epidemics in resource poor settings with limited public health and sanitary facilities.

An effective inactivated whole cell bivalent cholera vaccine against Vibrio cholerae O1 and O139 was produced and implemented for public health purposes in Vietnam since the 1990s. This bivalent vaccine has been found to be safe and to confer significant protection against El Tor cholera in both children and adults and has over the last decade being used in the Vietnam to protect against cholera. This vaccine has further been reformulated by the IVI to meet WHO requirements and is now being produced in WHO prequalified vaccine company in India.

The reformulated vaccine has been shown to be safe and immunogenic in Indian children as well as adults. A large Phase III study of the vaccine, has recently been carried out in Kolkata, India in over 120,000 participants aged from one year and above. Results of the study are encouraging and the vaccine gives over 60% protection against cholera. The vibriocidal antibody response rate was 80% in children and 53% in adults. Following this study, the vaccine, designated as ShanChol has been licensed in India in April 2009. The vaccine is now being marketed in India and is available at a cost affordable for developing country settings.

Objective: The aim of the proposed study is to assess if the orally administered, killed, bivalent whole-cell cholera vaccine, ShanChol will be safe and immunogenic in different age groups in Bangladesh in children and adults.

Study design: This will be a randomized, double blind, placebo-controlled study on a total of 330 subjects, 165 vaccine and 165 placebo recipients. The specific aims will be to determine: i) safety and determine adverse events if any (ii) determine immune responses.

Relevance: The study of ShanChol on Bangladeshi children and adults will be able to give information regarding the safety and immunogenicity of the vaccine in Bangladeshi subjects. This information will be important for proceeding with larger studies in Bangladesh and if proven useful for introduction the cholera vaccine in the country in the future.

DETAILED DESCRIPTION:
Adults as well as children, both males and females will be recruited in the study from the urban suburbs around Dhaka city in Mirpur where we have been conducting other epidemiological and vaccine related studies. The community will be informed by our field staffs and interested persons might be enrolled in the study on the basis of inclusion/exclusion criteria.

Part I- Adults- 18-45 years of age (n=110):

Since this oral bivalent whole-cell cholera vaccine has not been tested in Bangladesh before, the study will be carried out in 3 age groups, i.e. adults, followed by toddlers and younger children. These study participants will be recruited from the field site in Mirpur. For this purpose, 55 adults (18-45 year old) will be given 2 doses of the bivalent whole-cell cholera vaccine and 55 adults will be given placebo. Safety will be clinically monitored for side effects for 3 days after each dose of study agent by home visits. Participants will be randomized to receive either 2 doses of the vaccine or placebo, given 14 days apart.

Part II- Children 2-5 years (n=110):

If the vaccine is found safe in the adult study, it will be tested in the toddlers in the field consisting of 55 children in each group. The children will be clinically monitored for side effects for 3 days after each dose of vaccine.

Part III- Children 12-23 months (n=110):

Children in the field site will be recruited for the study and study carried out as described above.

Study procedure:

Each phase of the study (Part I onwards) will be completed and based on the development, and progress, the next phase will be initiated. If the vaccine is found to be without adverse effects on the adults it will be tested in the children, 2-5 years of age and followed by the younger age group 12-23 months of age. The results will be presented to the Data Safety Monitoring Board after completing the safety surveillance part of each phase of the study and before proceeding to the next study group.

Surveillance for side effects:

The safety of the study agents will be monitored after the intervention has been initiated. In the community, supervision will be carried out by the physician and the trained research assistants and adverse reactions including diarrhea, vomiting, nausea and other local and systemic reactions recorded. For the all three groups, 3 consecutive days after the each dose of study agent, the participants or their guardians will be interviewed for recall of symptoms by health workers. All side-effects will be recorded up to 28 days in reaction surveillance forms for local and systemic reactions. If any adverse event or serious adverse events notified within the study period field clinic will be available for reporting and possible management of the event. Reported symptoms other than appetite loss will be graded as mild (noticeable), moderate (affecting normal daily activities) or severe (suspending normal daily activities). A clinical record form will be used to record all clinical signs and symptoms. In case of serious adverse effects the data will be entered in a separate form . If required the study subject will be hospitalized at the Mirpur Treatment Center or the ICDDR,B Dhaka Hospital under supervision of the study physicians..

Safety endpoint and safety evaluation:

The primary end point for evaluating safety will be defined as the occurrence of any of the following diarrhoea, vomiting or abdominal cramps of at least moderate grade. Diarrhea will be defined as three or more loose or liquid stools in any 24-h period over the 3 day surveillance period.

STUDY INTERVENTION Vaccine Each dose of the vaccine contains whole cell inactivated heat killed and formalin killed bacteria consisting of 600 ELISA Units (EU) of lipopolysaccharide (LPS). It consists of formalin-killed V. cholerae Inaba, El Tor biotype (strain Phil 6973). It also contains 300 EU LPS of heat-killed V. cholerae Ogawa classical biotype (Cairo 50); 300 EU LPS of formalin killed V. cholerae Ogawa classical biotype (Cairo 50); 300 EU LPS of heat-killed V. cholerae Inaba, classical biotype (Cairo 48); and 600 EU LPS of formalin killed V. cholerae O139 (4260B) (9). The vaccine has no detectable cholera toxin. The study agents (Vaccine or placebo) is packaged as liquid formulations in 1.5-ml doses. The vaccine will be given in two doses separated by a two week interval and administered by oral syringe without a needle after which each participant will be offered water. No buffer will be co administered.

Placebo The placebo consists of heat-killed Escherichia coli K12 and is identical in appearance to the vaccine. This strain has been used for placebo related studies in previous oral vaccine clinical trials in Bangladesh and elsewhere.

Random Allocation Eligible participants will be assigned to receive the vaccine or placebo in a 1:1 ratio according to the randomization schedule. Individual randomization lists for adults, toddlers and infants will be generated by statistician in IVI who will not involved in the study in any way.

The study agents will be labeled by different letter codes for three different phases at Shantha Biotechnics according to the list provided by IVI.

The field staff will allocate the study agents to the participants according to the next available number on entry into the trial which will be linked with the randomization list provided by IVI.

The randomization list will contain sequential numbers unique to each participant, and the block randomization (fixed block length of 4) process will be employed to ensure an effective balance between the interventions.

Data Safety Monitoring Board (DSMB):

A 4-5 member data safety and monitoring board (DSMB) will be formulated for this study by the Ethical Review Committee (ERC) of ICDDR,B. This will be comprised of members of the ERC, staff members of ICDDR,B and individuals from other institutions in Bangladesh. The team will also comprise an International member. The members will not be involved in the study in any way.

Blinding and Code Breaking Procedures Vials will be labeled by letter codes at Shanta Biotechnics according to the list provided by IVI. All study personnel and participants will be blinded to treatment assignment during the duration of the study.

The identity of the study agent will not be known to the participant or their parent/guardian, nor to personnel involved in the conduct or monitoring of the trial, such as investigators, study nurses/personnel before the completion of the study.

The PI will hold the sealed randomization list for use if necessary in case of adverse events that may be seen in the study by the DSMB. Otherwise the list will not be unblinded until completion of the study, and complete entry and editing of relevant data before initiation of the analyses. The entire data set will be locked prior to unblinding. If the intervention assignment is un-blinded due to any reason, the DSMB will be notified within 24 hours.

Subject withdrawal during the study Respective participants or parents of participating children may discontinue his/her participation at any time after enrollment without providing any reason. No replacement will occur for such withdrawals.

The following criteria should be checked at each visit subsequent to the intake of study agent

1. Use of any immunosuppressive or immune-modifying drugs during the study period (for corticosteroids this would mean ≥0.5 mg/kg.day)
2. Administration of immunoglobulins or any blood product during the study period If any of the above occurs that might compromise per protocol assessment (PP); however, they will not be withdrawn from the study and their data will be used in an "intention to treat" (ITT) analysis. The investigator(s) might also withdraw a participant if, in his/her clinical opinion, that is in the best interest of the participant concerned or if it is considered to be non-compliant with the protocol. A participant might also be withdrawn due to protocol violation, death or early termination of the study by the sponsor. Wherever possible, the tests and evaluations at termination visit, as specified in the protocol, will be carried out.

   Duration of the study period for individual participants The participants will remain in the study for up to 28 days.

   Schedule and description of observations and visits:

   The following schedule will be used in the study and the case report forms will be completed on each study day:
3. Day 0: After describing the study and initial verbal consent, medical history will be obtained and a thorough physical examination will be performed by a physician that will include measurement of the vitals signs. Once all eligibility criteria are met,the participant and in case of children the parent will be asked to sign the informed consent form. A blood and stool sample would be collected for determining the baseline immunological assay for immune responses. Following this, the participant will be allocated to the study intervention according to the randomization list (vaccine or placebo). Voluntary and solicited reactogenicity will be assessed symptoms and immediate adverse events recorded with 1 h of intake of the study agent. The participants will then be allowed to go home
4. Day 1: Participants return to the study center to be monitored for voluntary and solicited symptoms and adverse events.
5. Day 2: Participants will return to the study centre or will be visited at home (in exceptional circumstances, when parents cannot bring the participant to the study centre) to monitor for voluntary and solicited symptoms and adverse events.
6. Day 7: (up to +3 days): Participants return to the study center. Blood sample will be collected at clinic and stool sample will be collected from home or at clinic for testing of vaccine specific immunologic responses in study participants.
7. Day 14: (± 2 days): Participants return to the study center. The participant will be allocated to the study intervention for second time according to the randomization list (vaccine or placebo).by a blinded third party dispenser.
8. Day 14-16: Participants return to the study centre or will be visited at home (in exceptional circumstances, when parents cannot bring the participant to the study centre) to monitor for voluntary and solicited symptoms and adverse events. Voluntary and solicited reactogenicity will be assessed symptoms and immediate adverse events.
9. Day 21: (± 3 days) Blood and stool will be sampled for testing of vaccine specific post immunization response.
10. Day 28: (± 3 days) Clinical evaluation and Study Termination Sample Size Calculation and Outcome (Primary and Secondary) Variable(s) Safety and Immunogenicity study of the Shantha cholera vaccine: The ''non-inferiority'' approach using a 1 -sided 95% confidence interval was used to calculate the sample size since this allowed us to rule out clinically unacceptable high rates of diarrheal adverse event occurring during the 3 days after either dose as well as establish that the vaccine induced adequate seroconversion to V. cholerae O1 among recipients. Assuming a 10% diarrheal rate among placebo and vaccine recipients alike, to exclude a vaccine-placebo difference in the rate of diarrhea of greater than 20% (upper boundary of the 1-tailed 95% confidence interval) with a power of 0.9, the minimum number of subjects required for each group was in each group for both adverse event was 46. The sample size is calculated with the assumptions that it is important to evaluate whether the vaccine induces acceptable serum vibriocidal responses in relation to the placebo group. Based on an immunogenicity study of the whole-cell killed oral cholera vaccine in Bangladesh, we make the following assumptions. For serum vibriocidal responses, defined as >4-fold increases between baseline and post-second dose in either Inaba or Ogawa antibodies, for each age group (12-23 months, 2-5 years and 18-45 years), we assume 1) the background rate of responses in the placebo group will be 5% after the second dose and 2) the true rate of vibriocidal responses in the vaccine groups is 25%. At p <0.05 (1-tailed), 0.8 power, and a 1 to 1 allocation of vaccine and placebo, a total of 46 subjects per group would be needed. Thus for safety and immunological responses the number is 46 per group. With 15% attrition rate, it is 53. We will select 55 in each group (110 per age group for both vaccine and placebo recipient).

We will, therefore, select 55 subjects per arm in each age group, with a total of 330 subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 12-23 months for younger children group, 2-5 years for the toddler group and 18-45 years for the adult group.
2. Sex: Either
3. Consent: Written informed consent from study participants and parents in case of children.
4. Compliance to study procedures: e.g. available for follow-up visits and agrees to specimen collection.
5. Apparently healthy: as determined by medical history, physical examination findings, and clinical judgment of the study physician.

Exclusion Criteria:

1. Chronic disease: history or evidence of chronic illness.
2. Gastrointestinal symptoms such as abdominal pain or cramps, loss of appetite, nausea, general ill-feeling or vomiting in the past 24 hours or abdominal pain lasting for more than 2 weeks in the past 6 months
3. Intake of any anti-diarrheal medicine or antimicrobial therapy the past week.
4. Acute disease one week prior to enrollment, with or without fever ≥38ºC .
5. Receiving of cholera vaccine any time in the past, and any other live or killed enteric vaccine in the last 4 weeks.
6. Diarrhea within 6 week period at screening.

Ages: 12 Months to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 330 (Actual)
Dates: Start 2010-01; Primary Completion 2010-08 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Safety and Reactogenicity: of orally administered killed, bivalent whole-cell cholera vaccine cholera vaccine, ShanChol | 1 year

SECONDARY OUTCOMES:
Immunogenicity: of cholera vaccine assessed by serum vibriocidal antibody responses as well as serological and mucosal responses to vaccine antigens and compare it with those obtained with placebo recipients. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Firdausi Qadri, PhD, Principal Investigator — International Centre for Diarrhoeal Disease Research, Bangladesh
Locations (1):
- Dr. Firdausi Qadri, Mirpur, Dhaka, Bangladesh

REFERENCES:
- [Background] Sur D, Lopez AL, Kanungo S, Paisley A, Manna B, Ali M, Niyogi SK, Park JK, Sarkar B, Puri MK, Kim DR, Deen JL, Holmgren J, Carbis R, Rao R, Nguyen TV, Donner A, Ganguly NK, Nair GB, Bhattacharya SK, Clemens JD. Efficacy and safety of a modified killed-whole-cell oral cholera vaccine in India: an interim analysis of a cluster-randomised, double-blind, placebo-controlled trial. Lancet. 2009 Nov 14;374(9702):1694-702. doi: 10.1016/S0140-6736(09)61297-6. Epub 2009 Oct 8. PMID 19819004
- [Background] Kanungo S, Paisley A, Lopez AL, Bhattacharya M, Manna B, Kim DR, Han SH, Attridge S, Carbis R, Rao R, Holmgren J, Clemens JD, Sur D. Immune responses following one and two doses of the reformulated, bivalent, killed, whole-cell, oral cholera vaccine among adults and children in Kolkata, India: a randomized, placebo-controlled trial. Vaccine. 2009 Nov 16;27(49):6887-93. doi: 10.1016/j.vaccine.2009.09.008. Epub 2009 Sep 15. PMID 19761838
- [Background] Mahalanabis D, Lopez AL, Sur D, Deen J, Manna B, Kanungo S, von Seidlein L, Carbis R, Han SH, Shin SH, Attridge S, Rao R, Holmgren J, Clemens J, Bhattacharya SK. A randomized, placebo-controlled trial of the bivalent killed, whole-cell, oral cholera vaccine in adults and children in a cholera endemic area in Kolkata, India. PLoS One. 2008 Jun 4;3(6):e2323. doi: 10.1371/journal.pone.0002323. PMID 18523643